CLINICAL TRIAL: NCT05064969
Title: A Blended Intervention Based on Acceptance and Commitment Therapy (ACT) for Informal Caregivers of People With Dementia- A Mixed-method Approach to Evaluate Feasibility, Acceptability and Preliminary Effectiveness
Brief Title: Acceptance and Commitment Therapy for Informal Caregivers of People With Dementia
Acronym: ACT-IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NL77389.068.21
Record Dates: First submitted 2021-09-03; First posted 2021-10-01 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: No Specific Conditions
Keywords: Acceptance and Commitment Therapy; Informal caregivers; Internet-based intervention; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm non-randomised (Experimental): This study includes a baseline assessment, a 9-week (with the possibility of extension to 12 weeks) blended intervention period, a post-intervention assessment, and two follow-ups at 3 and 6 months. Informal caregivers of people with dementia (with at least 18-year-old) with no restriction in terms of sex, educational level, or ethnic background will be included.
  Interventions: Behavioral: Blended intervention based in acceptance and commitment therapy

INTERVENTIONS:
Behavioral: Blended intervention based in acceptance and commitment therapy — Blended intervention includes completing 9 e-modules consist of written material, videos, and assignments (one e-module per week) that can be completed over 9 to 12 weeks AND 9 (to 12 ) coaching sessions (telephone call). Weekly coaching will be offered by a motivational coach based in Maastricht University.
  After the post-intervention assessments, individuals will receive monthly calls from the motivational coach as "booster sessions". Booster sessions will be received on monthly basis for a period of 6 months (one session per month) and until the last follow-up assessment. Communication with participants will take place online or via telephone.

SUMMARY:
Dementia has a major impact on people with dementia and their family. Informal caregivers of people with dementia are at higher risk of developing depressive symptoms compared to informal caregivers of people with other chronic diseases. Therefore, supporting this group of informal caregivers is particularly important. With an online program based on Acceptance and Commitment Therapy (ACT), this study supports caregivers of people with dementia to lead a more meaningful and less stressful life. In addition to following the online program, caregivers are supported weekly by a coach, who helps to set goals, map important values in life, and take actions in relevant areas. The current study aims to examine the (1) feasibility and acceptability of the intervention and its procedure and; (2) preliminary effectiveness of the intervention on clinical outcomes (e.g. psychological flexibility and self-competence); and (3) maintenance of change after the intervention in short-and long-term follow-ups. This study includes a single-arm, non-randomized trial with a baseline assessment, a 9-week internet-based intervention period, a post-intervention assessment, and two follow-ups at 3 and 6 months. ACT is a promising form of therapy that has previously been shown to be effective in increasing the mental well-being of caregivers. However, this is the first study to combine online ACT modules, goal-setting, and weekly coaching for informal caregivers of people with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Adult informal caregivers (at least 18 years old)
* Access to the internet and having a tablet or computer
* Self-identified primary informal caregiver of a person diagnosed with dementia
* Taking care of the care recipient at least once a week for a period of at least three months
* Obtained informed consent *General (psychological) support from case managers will not count as professional psychological support, and therefore, informal caregivers who receive support from the case managers will also be included.

Exclusion Criteria:

* Caregivers who report having a cognitive disorder in their clinical record will be excluded (based on self-report).
* Caregivers who receive psychotherapy or psychopharmacological treatment within the last 3 months will be excluded (based on self-report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Assessing change in depression, anxiety, and stress | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention..
  Measure the emotional states of depression, anxiety and stress will be assessed by DASS-21 self-report questionnaire. DASS-21 has three sections (7-items per section) that measure depression, anxiety, and stress on a 4-point Likert scale (0= the statement did not apply to me at all, 4= the statement applied to me very much or most of the time. DASS-21 is a validated scale that has been used in previous studies and has been recommended for measuring the dimensions of depression, anxiety, and stress.
Assessing change in sense of competence | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention..
  Informal caregivers' sense of competence indicates the feelings of being capable of caring for a person with dementia. Short Sense of Competence Questionnaire (SSCQ) is a valid and reliable scale which has been used in previous studies with a similar target population and consists of seven items rated on a 5-point scale from 1 ("agree very strongly") to 5 ("disagree very strongly")
Assessing change in self efficacy | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention..
  The Caregiver Self-Efficacy Scale (CSES) is based on a Dutch adaptation of the Lorig et al. CSES evaluates caregiver self-efficacy (four item) and service-use self-efficacy (five items) and item scores range from 1 (uncertain) to 10 (very certain). Previous research has shown that CSES is valid and reliable
Assessing change in perceived burden | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention..
  Caregiver burden will be measured by a one-item questionnaire. The perseverance-time question will ask: if the informal caregiver's current situation persists, for how long (in month) the informal caregiver thinks they are able to maintain caregiving. This questionnaire is a good predictor for institutionalisation.
Acceptability | Will be assessed after completing the 9-week intervention
  Will be assessed qualitatively during a semi-structured interview based on Program Participation Questionnaire (PPQ)
Perceived feasibility | Will be assessed after completing each module (during the intervention). 9 time for 9 modules.
  Brief self-report feasibility questionnaire
Perceived feasibility and acceptability | After the last follow up assessment (6-month)
  Will be assessed qualitatively during the semi-structured interview
Attrition | During the study (duration of study is expected to be 1.5 year)
  Number of drop outs of study after collecting informed consent
Perceived feasibility and acceptability | 9 (to 12) times. One telephone call per week over 9 (to 12) weeks of intervention.
  Will be assessed qualitatively during coaching sessions

OTHER OUTCOMES:
Assessing change in psychological flexibility | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention.
  Psychological flexibility is defined as the ability to be accepting, flexible and conscious in facing challenging situations and the ability to stay engaged with valued activities. This factor will be assessed by Acceptance and Action Questionnaire II, (AAQ-II) which has been reported to be valid, reliable and psychometrically consistent . 10 Items are scored on a 7-point Likert scale and higher scores indicate more psychological flexibility
Assessing change in resilience | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention.
  Changes in psychological flexibility and functional coping with negative thoughts and feelings in informal caregivers will be assessed using the Flexibility Index Test (FIT-60). This reliable and valid questionnaire will assess six different ACT processes (acceptance, diffusion, self as context, attention to present moment and values, and dedicated action) and can monitor the progress of the ACT therapy. The questionnaire consists of 60 items and is scored on a seven-point Likert scale (0= completely disagree, 6= completely agree). Higher score reflects on higher psychological flexibility.
Assessing change in values | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention.
  Important areas of life will be identified by the Valued Living Questionnaire (VLQ), which individuals rate level of importance of 12 different areas (e.g. family, work) on 10-point Likert scale (1= the area is not important at all, 10= the area is very important). The most important area will be considered as individuals' "value" at their current stage of life. The psychometric properties have been investigated in previous studies.
Assessing change in committed actions | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention.
  The extent to which individuals have been actively living in accordance with their values will be assessed by the Engaged Living Scale (ELS). ELS has been recommended for assessing committed actions and value engagement . ELS consists of 16-items in which individual should reflect in statements based on 5-point Likert scale (1=strongly disagree, 5= strongly agree)
Assessing change in gaol attainment | Will be assessed at baseline, after completing the intervention (9 to 12 weeks), 3month after intervention, and 6 month after intervention.
  Goal-attainment scaling will be conducted qualitatively and will be measured as part of the weekly coaching and booster sessions. Level of goal achievement since the last coaching session and the extent to which participants could achieve their goals at expected level will be discussed

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Dara will be shared and handled based on the data management plan supported by the Clinical Trial Centre Maastricht.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Atefi GL, van Knippenberg RJM, Bartels SL, Verhey FR, de Vugt M. Blended intervention based on acceptance and commitment therapy for informal caregivers of people with dementia (ACT-IC): protocol of a mixed-methods feasibility study. BMJ Open. 2023 Sep 13;13(9):e070499. doi: 10.1136/bmjopen-2022-070499. PMID 37709305